CLINICAL TRIAL: NCT01653886
Title: Palatability of Meals That Vary in Fat and Energy Density. A Pilot Study to the Behavioral Response to Short-Term (Two Day) Positive Energy Balance Through Overfeeding (ENERGY I)
Brief Title: Palatability (Energy I Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: PBRC 10017-P
Record Dates: First submitted 2012-07-26; First posted 2012-07-31 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Energy Density
Keywords: Palatability; Taste
MeSH Terms: interventions — Breakfast; Lunch; Meals

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pilot Group 1 (Experimental): Each Participant completed taste tests at breakfast, lunch and dinner consisting of the 4 menus (baseline, high fat-high energy density, high fat-low energy density, and high carbohydrate-low energy density).
  Interventions: Other: Breakfast (1-2 hours, in the morning); Other: Lunch (1-2 Hours, at midday); Other: Dinner (1-2 hours, in the afternoon)
- Pilot Group 2 (Experimental): Each Participant completed taste tests at breakfast, lunch and dinner consisting of the 4 menus (baseline, high fat-high energy density, high fat-low energy density, and high carbohydrate-low energy density).
  Interventions: Other: Breakfast (1-2 hours, in the morning); Other: Lunch (1-2 Hours, at midday); Other: Dinner (1-2 hours, in the afternoon)
- Pilot Group 3 (Experimental): Each Participant completed taste tests at breakfast, lunch and dinner consisting of the 4 menus (baseline, high fat-high energy density, high fat-low energy density, and high carbohydrate-low energy density).
  Interventions: Other: Breakfast (1-2 hours, in the morning); Other: Lunch (1-2 Hours, at midday); Other: Dinner (1-2 hours, in the afternoon)
- Pilot Group 4 (Experimental): Each Participant completed taste tests at breakfast, lunch and dinner consisting of the 4 menus (baseline, high fat-high energy density, high fat-low energy density, and high carbohydrate-low energy density).
  Interventions: Other: Breakfast (1-2 hours, in the morning); Other: Lunch (1-2 Hours, at midday); Other: Dinner (1-2 hours, in the afternoon)

INTERVENTIONS:
Other: Breakfast (1-2 hours, in the morning) — You will be required to taste small portions (1 to 2 bites) of 4 different breakfast meals. You will be asked to reate the taste after each meal. Meals will vary in fat and energy density, and will consist of two high fat diets and a high carbohydrate diet. Energy density is the ammount of enregy of kilocalories in one gram of the food.
Other: Lunch (1-2 Hours, at midday) — You will be required to taste small portions of 4 different lunch meals. You will be asked to reate the taste after each meal. Meals will vary in fat and energy density, and will consist of two high fat diets and a high carbohydrate diet. Energy densityis the ammount of enregy of kilocalories in one gram of the food.
Other: Dinner (1-2 hours, in the afternoon) — You will be required to taste small portions of 4 different dinner meals. You will be asked to reate the taste after each meal. Meals will vary in fat and energy density, and will consist of two high fat diets and a high carbohydrate diet. Energy densityis the ammount of enregy of kilocalories in one gram of the food.

SUMMARY:
A pilot study was conducted to develop the study menus that were similar in appearance, aroma, and taste.

DETAILED DESCRIPTION:
The aim of the pilot study was to test for differences in palatability ratings of the four menus that will be administered during the ENERGY I project. During the pilot study, palatability ratings were collected for each meal (breakfast, lunch, and dinner) from four different menus that were served to participants during the main ENERGY I trial. The menus consist of three diets that vary in dietary fat and energy density: 1) high fat/high energy density, 2) high fat/low energy density, and 3) high carbohydrate/low energy density. In addition to these three menus, the menu from the baseline period of the trial will also be tested for palatability.

ELIGIBILITY:
Inclusion Criteria:

* You are between the ages of 18 and 50, inclusive, if you are a male or between the ages of 18 and 45, inclusive, if you are a female.
* your body mass index (BMI) is between 25 and 30 kg/m2, inclusive
* For females, if you have regular menstrual periods, with no less than 28 day cycles.

Exclusion Criteria:

* you have a chronic disease that affects body weight, appetite, or metabolism, such as diabetes and cardiovascular disease.
* You use prescriptions or over-the-counter medications or herbal products that affect metabolism or body weight (e.g. weight loss medications such as sibutramine, or orlistat).
* You have symptoms of depression or excessive dietary restraint.
* You have an allergy to one or more of the test foods.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Palatability | 2 days
  The aim of the study is to test for differences in palatability rats of four menus that will be administered during the ENERGY I project. During the pilot study, weill will collect palatability ratings for each menu (breakfast, lunch, and dinner) from four different menus that will be served to participants during the main trial. The menus consist of three diets and baseline. that vary in dietary fat and energy density : 1) high fat/high energy density, 2) hgih fat/low energy density, and 3) high carbohydrate/low energy density.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Apolzan JW, Bray GA, Hamilton MT, Zderic TW, Han H, Champagne CM, Shepard D, Martin CK. Short-term overeating results in incomplete energy intake compensation regardless of energy density or macronutrient composition. Obesity (Silver Spring). 2014 Jan;22(1):119-30. doi: 10.1002/oby.20587. Epub 2013 Sep 10. PMID 23913807